CLINICAL TRIAL: NCT05620901
Title: The Evaluation of the Safety and Efficacy of Sustained Release Dexamethasone Intracanalicular Insert (DEXTENZA) in Pediatric Patients Following Retinal Surgery or Laser Treatment Under Anesthesia (TENDER)
Brief Title: DEXTENZA in Pediatric Patients Following Retinal Surgery or Laser Treatment Under Anesthesia
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Lejla Vajzovic, MD, FASRS (Other)
Responsible Party: Sponsor-Investigator, Lejla Vajzovic, MD, FASRS, Principal Investigator, Duke University
Organization: Duke University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00107533
Record Dates: First submitted 2022-11-10; First posted 2022-11-17 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-01

CONDITIONS: Vitreoretinopathy; Coats' Disease; Exudative Retinopathy; Lattice Degeneration; Retinal Hole; Sickler's Syndrome; Retinal Detachment Rhegmatogenous; Retinal Detachment Exudative; Retinal Detachment Traction
MeSH Terms: conditions — Retinal Telangiectasis; Retinal Perforations | interventions — Calcium Dobesilate; prednisolone acetate

STUDY DESIGN:
Intervention Model Description: The study aims to enroll 30 pediatric patients undergoing routine retinal surgery or laser treatment under anesthesia. Patients in each treatment group (surgery or laser) will be randomized 2:1 at the time of surgery/ laser to receive either the Dextenza insert or the Control (Prednisolone Acetate 1%) steroid drops tapered for 28 days post-operatively.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment Arm (Experimental): Dextenza insert intraoperatively for perioperative ocular inflammation and pain. These patients will not be prescribed topical steroid drops post-operatively
  Interventions: Drug: Dextenza 0.4Mg Ophthalmic Insert
- Control Arm (Active Comparator): Prednisolone forte 1% steroid drop taper for 28 days post-operatively to treat perioperative ocular inflammation and pain; drops four times per day (QUID) on days 0-7, three times per day (TID) on days 7-14, twice per day (BID) on days 14-21 and once per day (QD) on days 21-28.
  Interventions: Drug: Pred Forte

INTERVENTIONS:
Drug: Dextenza 0.4Mg Ophthalmic Insert — DEXTENZA (dexamethasone ophthalmic insert) 0.4 mg, for intracanalicular use
  Arms: Treatment Arm
Drug: Pred Forte — To treat perioperative ocular inflammation and pain;
  Arms: Control Arm

SUMMARY:
The Tender Study is a prospective, open-label, single-center, randomized, investigator-initiated clinical study seeks to investigate the safety and efficacy of the DEXTENZA insert in pediatric patients following retinal surgery or laser treatment under anesthesia.

DETAILED DESCRIPTION:
The study aims to enroll 30 pediatric patients undergoing routine retinal surgery or laser treatment under anesthesia. Patients in each treatment group (surgery or laser) will be randomized 2:1 at the time of surgery/laser to receive either:

1. Treatment Arm: Dextenza insert intraoperatively for perioperative ocular inflammation and pain. These patients will not be prescribed topical steroid drops post-operatively, or
2. Control Arm: Prednisolone forte 1% steroid drop taper for 28 days post-operatively to treat perioperative ocular inflammation and pain; drops four times per day (QUID) on days 0-7, three times per day (TID) on days 7-14, twice per day (BID) on days 14-21 and once per day (QD) on days 21-28.

Each treatment group (surgery or laser) will include 15 patients total, 10 receiving Dextenza and 5 receiving the control drug. Drops for dilation and antibiotic coverage will be used as clinically indicated in all groups throughout the study period. Follow up will occur at post-op day 1, 7, 28/30 and 45 ( +/- three days for all post-operative timepoints).

ELIGIBILITY:
Inclusion Criteria:

Pediatric patients undergoing routine retinal surgery or laser treatment under anesthesia for a variety of visual conditions. These conditions and procedures include but are not limited to:

Conditions:

* Familial Exudative Vitreoretinopathy
* Coats' Disease
* Exudative Retinopathy
* Lattice degeneration
* Retinal holes
* Sickler's syndrome
* Retinal detachment, rhegmatogenous
* Retinal detachment, exudative
* Retinal detachment, tractional

Procedures

* Laser photocoagulation
* Cryotherapy
* Retinal detachment repair with scleral buckle and cryotherapy
* Retinal detachment repair with vitrectomy
* Written informed consent from parent/legal guardian

Exclusion Criteria:

Preprocedural

* Active or history of chronic or recurrent inflammatory eye disease in either eye
* Any patient of reproductive potential that has a positive pregnancy test during pre-procedural testing
* Active or history of increased ocular pressure
* Patients with active corneal, conjunctival, and canalicular infections
* Patients with punctal stenosis or other punctal anatomical abnormalities that would not be conducive with device insertion
* Nasolacrimal duct obstruction
* Laser or incisional ocular surgery during the study period and 6 months prior in the study eye
* current use of systemic or topical steroids or NSAIDS on a regular basis
* History of autoimmune disease that may interfere with treatment/outcomes
* Ocular pain at the time of screening
* Known malignancy
* Current use of cyclosporin or a TNF blocker
* Ocular hypertension IOP >25, actively taking medications for ocular hypertension, any history of IOP spikes in either including steroid associated IOP elevation
* Congenital ocular lid and tear duct system abnormalities (e.g. congenital ectropion/entropion, trichiasis)
* Evidence of acute external ocular infection of the study eye
* Active or history of HSV
* Previous trauma causing deformity
* Previous enrollment or current enrollment with another clinical trial within the last 30 days that may interfere with treatment
* Known allergies to product under investigation
* Inability to engage in VA testing
* Investigator determines that the candidate is not eligible for participation based on clinical or historical factors that would interfere with treatment or impact patient safety not specified above
* Current artificial tear use >4x daily
* Current use of any topical ocular drops
* Anyone who, in the opinion of the investigator, would not be a good candidate for the study.

Intraoperatively

* Multiple procedures required
* Complication occurs that surgeon determines makes the patient ineligible for study inclusion
* Unsuccessful dilation of the punctum to 0.7mm when dilation attempted
* during the exam under anesthesia, if it is decided that periocular Kenalog injection is indicated this patient fails screen and will no longer be eligible for the study

Ages: 3 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 16 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2025-02-11 (Actual); Study Completion 2025-02-24 (Actual)

PRIMARY OUTCOMES:
Pain as measured by the FLACC pain scale | up to Day 45 post-op
  The Face, Legs, Activity, Cry and Consolability (FLACC) scale is an observational scale. comprised five behavioural indicators that are scored from zero to two. The pain score is the sum of the item scores and ranges from zero to 10. A lower score indicates minimal to no pain while high scores indicate moderate to severe discomfort.

SECONDARY OUTCOMES:
Incidence of adverse events | up to Day 45 post-op
  Adverse events are addressed/ assessed at each visit
Severity of Adverse Events | up to Day 45 post-op
  Adverse events are addressed/ assessed at each visit
Degree of inflammation (AC cell count) | up to Day 45 post-op
  Inflammation is evaluated at each visit during the slit lamp and fundus exam as measured by the ocular inflammation grading scale
Resolution of inflammation or less cell on follow up post op exams | up to Day 45 post-op
  Inflammation is evaluated during slit lamp and fundus exams during each post-op visit
Resolution of pain | up to Day 45 post-op
  This will be measured by using the FLACC Pain Rating Scale. The Face, Legs, Activity, Cry and Consolability (FLACC) scale is an observational scale comprised five behavioural indicators that are scored from zero to two. The pain score is the sum of the item scores and ranges from zero to 10
Ratio of Intraocular pressure increase with insert | up to Day 45 post-op
  Intraocular pressure is assessed at each visit
Percentage of patients with rebound inflammation from baseline through post-op care | up to Day 45 post-op
  Level of inflammation is evaluated at each post-op visit during slip lamp and fundus exams
Percentage of patients that were given supplementary prednisolone drops | up to Day 45 post-op
  Supplemental treatment and additional drops needed will be documented at each subsequent visit
The number of drops needed in these patients | up to Day 45 post-op
  Supplemental treatment and additional drops needed will be documented at each subsequent visit
Mean change in Best Corrected Visual Assessment (BCVA) | up to Day 45 post-op
  Determined by using either ETDRS or HOTV chart testing depending on age.
Caregivers Treatment Adherence | up to Day 45 post-op
  Documented at each subsequent visits and with the primary caregiver satisfaction survey at Day 45. This is a subjective survey for each participants' family.

CONTACTS AND LOCATIONS:
Overall Officials: Lejla Vajzovic, MD, Principal Investigator — Duke Eye Center
Locations (1):
- Duke Eye Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No